CLINICAL TRIAL: NCT03162497
Title: Effect of Topical Azithromycin on Tear Film Thickness in Patients With Meibomian Gland Dysfunction - Comparison to Oral Treatment With Doxycycline
Brief Title: Effect of Topical Azithromycin on Tear Film Thickness in Patients With Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPHT-030815
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2022-04

CONDITIONS: Dry Eye Syndromes; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Azithromycin; Doxycycline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin (Experimental): Preservative-free azithromycin 15mg/g (Azyter® Augentropfen im Einzeldosisbehältnis, Thea, Clermont-Ferrand, France) one drop twice daily for two days then once daily for 26 days
  Interventions: Drug: Azithromycin
- Doxycycline (Active Comparator): Doxycycline 100mg (Doxycycline "Genericon", Genericon Pharma GmbH, Graz, Austria) twice daily for 6 weeks
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 15mg/g eyedrops
  Arms: Azithromycin
Drug: Doxycycline — Doxycycline 100 mg per os
  Arms: Doxycycline

SUMMARY:
Meibomian gland dysfunction (MGD) is among the leading causes for dry eye syndrome (DES), affecting millions of people worldwide. We have shown in a previous study that tear film thickness (TFT) is reduced in patients with DES and that this reduction correlates with tear break up time (BUT) as well as with the severity of subjective symptoms. Even though systemic tetracyclines as well as topical azithromycin can be used for the treatment of MGD, it seems that topical azithromycin is more effective than tetracyclines and also has the advantage of better tolerability. The hypothesis of the present study is that topical treatment with azithromycin leads to a more pronounced increase in TFT compared to oral doxycycline in patients with DES caused by MGD.

The objective of this study is to compare the effect of treatment with topical azithromycin or oral doxycycline on tear film thickness in patients with DES caused by MGD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Signs of meibomian gland plugging or expressibility of the meibomian glands.
* DES most likely caused by MGD, no other cause identifiable which is more likely (e.g. intake of concomitant medication that could induce DES, systemic diseases such as systemic arthritis or diabetes), as judged by the investigator
* Signed and dated written informed consent.
* History of dry eye syndrome for at least 3 months
* Normal ophthalmic findings except dry eye syndrome and MGD, ametropia < 6 Dpts
* BUT ≤ 10 seconds

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks before the screening visit
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Presence or history of a severe ocular condition that will interfere with the study aim as judged by the clinical investigator
* Treatment with corticosteroids in the 4 weeks preceding the study
* Wearing of contact lenses
* Topical treatment with any ophthalmic drug in the 4 weeks preceding the study except topical lubricants Ocular infection
* Ocular surgery in the 6 months preceding the study
* Pregnancy, planned pregnancy or lactating
* Contraindication against the use of topical azithromycin or oral doxycycline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Change in tear film thickness | 8 weeks
  Change in tear film thickness measured with high resolution OCT before, during and after treatment period.

SECONDARY OUTCOMES:
Change in lipid layer thickness | 8 weeks
  Change in lipid layer thickness measured with the Lipiview device before, during and after treatment period.
Change in break up time (BUT) | 8 weeks
  Change in tear break up time (BUT) measured with fluorescein before, during and after treatment period.
Change in Visual Acuity | 8 weeks
  Change in Visual Acuity assessed before, during and after treatment period.
Change in tear osmolarity | 8 weeks
  Change in tear osmolarity assessed before, during and after treatment period.
Change in Staining of the cornea with fluorescein | 8 weeks
  Change in Staining of the cornea with fluorescein assessed before, during and after treatment period.
Change in impression cytology | 8 weeks
  Change in impression cytology assessed before, during and after treatment period.
Change in Schirmer I test | 8 weeks
  Change in Schirmer I test assessed before, during and after treatment period.
Change in Subjective symptoms of dry eye syndrome (OSDI© questionnaire) | 8 weeks
  Change in Subjective symptoms of dry eye syndrome (OSDI© questionnaire) assessed before, during and after treatment period.
Change in intraocular pressure | 8 weeks
  Change in intraocular pressure assessed before, during and after treatment period.
Change in meibography | 8 weeks
  Change in meibography assessed before, during and after treatment period.
Change in conjuctival staining with lissamine green | 8 weeks
  Change in conjuctival staining with lissamine green assessed before, during and after treatment period.
Change in corneal sensitivity | 8 weeks
  Change in corneal sensitivity assessed before, during and after treatment period.
Change in signs and symptoms of meibomian gland disease (MGD) | 8 weeks
  Change in signs and symptoms of meibomian gland disease (MGD) assessed before, during and after treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Gerhard Garhofer, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schlatter A, Hommer N, Kallab M, Stegmann H, Zeller K, Palkovits S, Findl O, Werkmeister RM, Schmetterer L, Garhofer G, Schmidl D. Effect of Treatment with Topical Azithromycin or Oral Doxycycline on Tear Film Thickness in Patients with Meibomian Gland Dysfunction: A Randomized Controlled Trial. J Ocul Pharmacol Ther. 2023 Jul;39(6):371-378. doi: 10.1089/jop.2022.0186. Epub 2023 Jun 16. PMID 37327369